CLINICAL TRIAL: NCT02716337
Title: Target Versus Standard Human Milk Fortification in Very Low Birth Weight Preterm Infants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Prof. Pier Mannuccio Mannucci, PHD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Target HM fortification
Record Dates: First submitted 2016-03-07; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Postnatal Growth Failure of Preterm Infants; Human Milk Fortification
Keywords: human milk target fortification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Other): In the intervention group VLBW infants were fed target fortified human milk Growth and safety were compared to a historical group of VLBW infants fed with standard fortified human milk
  Interventions: Dietary Supplement: Addition of human milk fortifiers according to human milk analysis

INTERVENTIONS:
Dietary Supplement: Addition of human milk fortifiers according to human milk analysis

SUMMARY:
The prevention of postnatal growth failure in very low birth weight (VLBW) preterm infants is of utmost importance. Standard fortification is the most commonly used supplementation practice but it does not consider the native variability of human milk. Data on efficacy and safety of prolonged target fortification are scarce. The investigators performed a prospective interventional study in VLBW preterm infants, exclusively fed with human milk, to test efficacy and metabolic safety of target fortification in these preterm infants.

DETAILED DESCRIPTION:
The prevention of postnatal growth failure in very low birth weight (VLBW) preterm infants is of utmost importance. Fortified human milk is the goal for preterm infants' nutrition. Standard fortification is the most commonly used and safe supplementation practice but it does not consider the native variability of human milk. Data on efficacy and safety of prolonged target fortification are scarce. Prospective interventional study was conducted in VLBW preterm infants, exclusively fed with human milk. Twenty-four hour collected pools of human milk were analyzed and targeted human milk fortification was performed during hospitalization. Weekly growth and daily growth velocity were compared with that of an historical group of VLBW preterm infants that had received standard fortified human milk. Osmolality, metabolic and gastrointestinal tolerance were monitored.

ELIGIBILITY:
Inclusion criteria:

* Birth weight < 1500 grams
* Gestational age < 32 weeks
* Birth weight > 10th percentile according to Fenton' growth chart
* Exclusively breast feeding during the entire hospital stay

Exclusion criteria:

- Presence of congenital malformations that could affect growth (congenital diseases, chromosomal abnormalities, chronic lung disease, severe brain disease, severe metabolic, cardiac or gastrointestinal diseases)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Daily growth velocity (g/kg/day) | From the beginning of human milk fortification until the end of hospitalization (mean period of treatment 4-5 weeks)

SECONDARY OUTCOMES:
weekly weight increase (g/week) | From the beginning of human milk fortification until the end of hospitalization (mean period of treatment 4-5 weeks)
weekly length increase (cm/week) | From the beginning of human milk fortification until the end of hospitalization (mean period of treatment 4-5 weeks)
head circumference increase (cm/week) | From the beginning of human milk fortification until the end of hospitalization (mean period of treatment 4-5 weeks)

OTHER OUTCOMES:
osmolality of fortified human milk | From the beginning of human milk fortification until the end of hospitalization (mean period of treatment 4-5 weeks)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morlacchi L, Mallardi D, Gianni ML, Roggero P, Amato O, Piemontese P, Consonni D, Mosca F. Is targeted fortification of human breast milk an optimal nutrition strategy for preterm infants? An interventional study. J Transl Med. 2016 Jul 1;14(1):195. doi: 10.1186/s12967-016-0957-y. PMID 27370649